CLINICAL TRIAL: NCT00694421
Title: Gas Supply, Demand and Middle Ear Gas Balance: Specific Aim 2
Status: Completed | Type: Observational
Sponsor: Cuneyt M. Alper (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Cuneyt M. Alper, Director of Research, ENT Department of CHP, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: 0607007; P50DC007667 (NIH)
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Upper Respiratory Infection
Keywords: otitis; Eustachian tube; virus; Middle ear disease
MeSH Terms: conditions — Respiratory Tract Infections; Otitis; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: adults who participate in study, "Social and Psychological Risks for Infectious Disease" here at Children's Hospital of Pittsburgh
- 2: children 2-6 years who participate in "Role of Virus and Genetic Susceptibility" study here at Children's Hospital of Pittsburgh

SUMMARY:
This study will test the hypothesis that constitutionally poorer Eustachian tube function predisposes to middle-ear pathology during a viral upper respiratory infection.

DETAILED DESCRIPTION:
The most well supported immediate cause of Otitis media (OM) is a pre-existing or concurrent viral upper respiratory tract infection (vURI). However, not all vURI episodes cause OM and a variety of predisposing factors has been suggested to explain this selectivity. Based on our preliminary work using a model of experimental viral infections in adults, we hypothesize that the constitutional efficiency of the Eustachian tube (ET) to supply the middle ear (ME) with gas and thereby stabilize ME pressure at near ambient is a primary risk factor for OM during vURI. Here, we test the hypothesis that constitutionally poorer ET function (F) predisposes to ME pathology during a vURI. Specifically, we will use ETF testing protocols relevant to the pressure-chamber to evaluate constitutional ETF in ≈ 160 susceptible, adult volunteers who will be exposed to rhinovirus as part of our funded study entitled "Social and Psychological Risks for Infectious Disease" (PI: S. Cohen, PI: CHP subcontract: WJ Doyle) and document the ETF and ME responses to infection over a 5-day post-exposure, cloister period.

Also, using protocols relevant to the pressure-chamber, we will evaluate constitutional ETF in 80 children who will be enrolled into our funded study entitled "Role of Virus and Genetic Susceptibility in Otitis Media" (PI: CM Alper) and followed for vURI and OM from October through April. From both data sets, we will extract measures of ETF efficiency and determine using logistic regression with appropriate control variables (e.g. demographic data etc) if a single or combination of ETF variables predicts an abnormal ME response in rhinovirus infected adults or OM during a rhinovirus cold in children.

ELIGIBILITY:
Inclusion Criteria:

* Participating/participated in one of the two identified studies

Exclusion Criteria:

* No longer meet inclusion/exclusion criteria of parent studies

Ages: 2 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Membership in one of the two identified source populations
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Eustachian tube function | 3 months (adults), 6 months (children)

CONTACTS AND LOCATIONS:
Overall Officials: William J Doyle, PhD, Principal Investigator — University of Pittsburgh; J Douglas Swarts, PhD, Study Director — University of Pittsburgh
Locations (1):
- ENT Research Center Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No